CLINICAL TRIAL: NCT00243958
Title: Aluminum and Auditory Function in ESRD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461701003
Record Dates: First submitted 2005-10-23; First posted 2005-10-25 (Estimated); Last update posted 2005-10-25 (Estimated); Status verified 2005-10

CONDITIONS: End-Stage Renal Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Hearing impairment either clinical or subclinical is a characteristic of some renal disease patients. The hearing impairment could be result from specific etiologies or chronic renal failure itself. The causes of hearing impairment in renal disease patients ranged from drugs intoxication in both auditory and renal function, like gentamycin or isoniazid, congenital disease like Alport syndrome or other collagen-defective renal disease, or just aging related. End-stage renal disease (ESRD) patients are special in many parts to general population who have hearing impairment. First, inflammation in ESRD patients is well-documented, second, they suffered from various underlying diseases which auditory function was potentially impaired, third, they need to undergo renal replacement therapy either hemodialysis (HD) or peritoneal dialysis (PD) to maintain their life. Dialysis itself was found to be a cause of hearing impairment, too. The biochemical change and constitutive inflammation status are thought to be implicated in the pathogenesis of hearing impairment in ESRD patients. Aluminum (Al) is a well-documented heavy metal, which predisposes to Alzheimer's disease, dementia or some neurologic diseases. Al intoxication is very rare in general health population but elevated serum Al level is easily found in ESRD patients since they can not excrete Al by damaged kidneys and dialyzers. Inner ear per se is a neurologic tissue, so if serum Al level in ESRD patients has any association in their haring function needs to be studied.

ELIGIBILITY:
Inclusion Criteria:

ESRD patients and healthy volunteers, without history of occupational noise exposure, ear infection, ear surgery, active systemic infection, previous ototoxic drugs exposure or congenital hearing defect

Exclusion Criteria:

Unsuitable to undergo hearing test, with history of occupational noise exposure, ear infection, ear surgery, active systemic infection, previous ototoxic drugs exposure or congenital hearing defect

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2005-10

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-Dun Wu, MD. PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Yun-Lin Branch, Douliu, Yun-Lin, Taiwan